CLINICAL TRIAL: NCT01439542
Title: FASTR: Fairly Brief Androgen Suppression and Stereotactic Radiotherapy for High Risk Prostate Cancer
Acronym: FASTR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Higher then expected Gr3 GU/GI toxicity
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, George Rodrigues, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-11-220; FASTR (Other: Principal Investigator)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: High risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation; Drug: Luteinizing Hormone Releasing Hormone (LHRH) Agonist

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — Clinical Target Volume 1 (CTV1): 25 Gy to nodes in 5 fractions, 1 fraction per week
  Clinical Target Volume 2 (CTV2): 40 Gy to prostate and seminal vesicles in 5 fractions, 1 fraction per week
Drug: Luteinizing Hormone Releasing Hormone (LHRH) Agonist — 12 months (2x6 month depot) of androgen suppression with LHRH agonist

SUMMARY:
The purpose of this study is to examine the safety of a shorter course of radiation treatments combined with one year of androgen deprivation therapy. The study will test this treatment in men with high risk prostate cancer who have significant other illnesses or circumstances such that conventional long term radiotherapy and hormone therapy is not recommended by their physician or desired by the patient.

DETAILED DESCRIPTION:
Randomized controlled trials have established the improved efficacy (better biochemical control and disease free survival) of combined radical radiation (70-80Gy/7-8 weeks) combined with long term hormone therapy (2-3 years of adjuvant luteinizing hormone releasing hormone (LHRH) agonist) compared to a primary hormone therapy or radiotherapy alone in men with locally advanced/high risk disease. While this approach may be tolerable in fit individuals, this combination may not be well tolerated by frail individuals or those who live at a distance who may find it difficult to attend for 7 weeks of radiation due to travel considerations. Those individuals with co-morbidities such as diabetes, coronary artery disease or osteoporosis may have those conditions exacerbated by long term hormone therapy.

This pilot study will explore the combination of a stereotactic body radiotherapy (SBRT) approach (designed to be iso-effective for late effects for standard radiotherapy) combined with one year of LHRH agonist for older men with high risk disease who are less fit (Vulnerable Elderly Score > 3) or men unwilling to undertake conventionally fractionated therapy and three years of adjuvant hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* High risk prostate cancer:

  * clinical stage T3 (cT3) prostate cancer or
  * pre-treatment PSA > 20 or
  * Gleason score>8 on Trans-Rectal Ultrasound (TRUS) biopsy
* Score of > 3 on the Vulnerable Elderly Scale or refuses standard radiotherapy + androgen deprivation therapy
* No evidence of extra-prostatic disease on screening bone scan and Computed Tomography (CT) scan (non-contrast CT used for CT simulation acceptable)
* Signed written and voluntary informed consent provided.
* Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Age ≥ 18 years

Exclusion Criteria:

* Patients not meeting the eligibility criteria
* Prior pelvic radiotherapy or brachytherapy
* Use of anti-coagulation (low molecular weight heparin or Coumadin)
* History of inflammatory bowel disease, Crohn's disease, diverticulitis or collagen vascular disease (other than rheumatoid arthritis)
* Previous treatment for malignancy (other than basal or squamous cell skin cancer) within 3 years of prostate cancer diagnosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Toxicity | year 1 of follow-up
  Assessment of late genitourinary and gastrointestinal toxicity at 1 year as assessed by the Common Toxicity Criteria
Toxicity | year 2 of follow-up
  Assessment of late genitourinary amd gastrointestinal toxicity at 2 years as assessed by the Common Toxicity Criteria
Toxicity | year 3 of follow-up
  Assessment of late genitourinary and gastrointestinal toxicity at year 3 as assessed by the Common Toxicity Criteria

SECONDARY OUTCOMES:
Disease Free Survival | years 1, 2 and 3 of follow-up
  3 year disease free survival (defined by absence of clinical relapse and prostatic specific antigen (PSA) failure as per the ASTRO Phoenix definition
Quality of Life | years 1, 2, and 3 of follow-up
  Quality of life as assessed by the Prostate Cancer Radiotherapy questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute; George Rodrigues, MD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada

REFERENCES:
- [Derived] Bauman G, Ferguson M, Lock M, Chen J, Ahmad B, Venkatesan VM, Sexton T, D'Souza D, Loblaw A, Warner A, Rodrigues G. A Phase 1/2 Trial of Brief Androgen Suppression and Stereotactic Radiation Therapy (FASTR) for High-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):856-62. doi: 10.1016/j.ijrobp.2015.02.046. Epub 2015 Apr 30. PMID 25936597